CLINICAL TRIAL: NCT01009320
Title: The Potential Interference of Magnets From a Surgical Magnetic Drape With Cardiac Pacemakers
Status: Completed | Type: Observational
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Valerie Zaphiratos, Principal investigator, Maisonneuve-Rosemont Hospital
Other Study IDs: HMRvzaphi; 09051
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Cardiac Pacemaker, Artificial
Keywords: Pacemaker; Magnets; Drape; Ferrite; Magnetic field; Pacemaker interference

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pacemaker with magnets: Patients with pacemakers who will be tested for magnetic interference with a magnetic drape.

SUMMARY:
Magnetic fields may interfere with the function of cardiac pacemakers. A magnetic drape to hold surgical instruments is widely used in surgery. The use of this drape on pacemaker patients has not yet been tested. Our objective is to conduct a clinical study to evaluate the potential interference of the surgical magnetic drape on patients with cardiac pacemakers. We are testing the magnetic drape on forty patients in the pacemaker clinic. The totality of the drape is applied over the pacemaker and depending on the result, the drape is either folded in two over the pacemaker or the magnets are applied individually up to the totality of the drape, 70 magnets. Thereafter, the drape is pulled in increments of 3 cm caudally until the interference is ceased. Results are in process as we are presently actively recruiting.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac pacemaker

Exclusion Criteria:

* Unstable angina
* Hemodynamic instability
* Subjects whom the cardiologist believes are unsuitable for asynchronous pacing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Out-patient clinic
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Asynchronous pacing | Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Philippe Fortier, MD, FRCPC, Study Director — Maisonneuve-Rosemont hospital, University of Montreal; Valerie Zaphiratos, MD, Principal Investigator — Maisonneuve-Rosemont hospital, University of Montreal
Locations (1):
- Maisonneuve-Rosemont hospital, Montreal, Quebec, Canada